CLINICAL TRIAL: NCT03373916
Title: Effectiveness and Implementation of a Peer Mentorship Intervention (PREVAIL) to Reduce Suicide Attempts Among High-Risk Adults
Brief Title: Peer Mentorship to Reduce Suicide Attempts Among High-Risk Adults
Acronym: PREVAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Paul Pfeiffer, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00137787; 1R01MH115111-01 (NIH)
Record Dates: First submitted 2017-11-28; First posted 2017-12-14 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Suicidal Ideation
Keywords: Peer Mentorship; Psychiatric Hospitalization; Suicide Risk
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Mentorship intervention (PREVAIL) (Experimental): PREVAIL peer mentorship
  Interventions: Behavioral: Peer mentorship; Behavioral: Enhanced Usual Care
- Enhanced Usual Care (EUC) (Active Comparator): Enhanced Usual Care
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Peer mentorship — The PREVAIL intervention will be delivered by a Certified Peer Support Specialist (CPSS) or Peer Recovery Coach. Participants will select a Peer to work with based on brief personal descriptions. Sessions may occur in-person (public place, the participant's home, or a research clinic space) or remotely (phone or video call). The first meeting will occur while the participant is hospitalized, and subsequent sessions will be scheduled per the participant's preferences, with a suggested frequency of twice weekly for weeks 1-2, weekly for weeks 3-8, and every other week for the last month. Sessions will last 1 hour on average and will consist of semi-structured conversations focused on protective factors such as hope, safety planning, and coping skills. Session structure and content are intentionally flexible to allow for general supportive listening, validation, sharing, and genuineness in the relationship, thereby increasing acceptability and implicit belongingness.
  Other Names: PREVAIL
  Arms: Peer Mentorship intervention (PREVAIL)
Behavioral: Enhanced Usual Care — The EUC condition will consist of a "caring message" from the study team via e-mail or text message (based on the participant's preference) 24-72 hours after discharge. An example message is, "We hope things are going well for you since you left the hospital. If you wish to reply, we'd be glad to hear from you." A list of local mental health resources will be available if participants reply and during the 3 and 6-month follow-up assessments. The EUC condition is modeled on prior studies of caring letters and brief contacts by health professionals after suicidal crisis and national recommendations to provide post-crisis follow-up contacts.
  Other Names: EUC

SUMMARY:
This is a single-blind, randomized controlled trial to test the effectiveness of a peer mentorship intervention (PREVAIL) for reducing suicide risk compared to enhanced usual care among participants (N=455) at high-risk for suicide recruited from inpatient psychiatric units.

DETAILED DESCRIPTION:
Amid consistently worsening suicide rates, in 2012 the U.S. Surgeon General's National Strategy for Suicide Prevention proposed to "change the narrative" about suicide prevention to include a focus on promoting hope and belongingness. Despite hopelessness and thwarted belongingness being among the most replicated risk factors for suicide, many widely implemented suicide prevention efforts instead emphasize the identification of acute suicide risk and referral to mental health treatment services. However, there are very few health service interventions known to reduce suicides among those identified as high risk. Those interventions shown to be effective have not achieved the wide scale implementation necessary to alter the trend of increasing suicide deaths. New interventions are needed, and one promising, scalable intervention with a novel approach to addressing the risk factors advocated by the Surgeon General is peer mentorship. A peer mentorship intervention, PREVAIL, has been piloted in a two-site randomized controlled trial (N=70) and is acceptable and feasible with enrollment of nearly half of eligible high-risk patients, mean completion of over 6 mentorship sessions, and 85% of sessions meeting fidelity standards for addressing the intended targets of hope and belongingness.

The aims of this hybrid effectiveness-implementation study are:

Specific Aim 1: Determine the effectiveness of the PREVAIL peer mentorship intervention for reducing suicide attempts and suicidal ideation among recently hospitalized adult psychiatric patients at high risk for suicide.

Specific Aim 2: Examine the mechanisms of peer mentorship by measuring the effects of PREVAIL on potential mediators,including hope and belongingness.

Specific Aim 3: Identify barriers and facilitators to implementation of PREVAIL.

ELIGIBILITY:
Inclusion Criteria:

1. are age 18 years or older,
2. are currently admitted to an inpatient psychiatric unit and have medical record documentation of suicidal ideation or suicide attempt at the time of admission,
3. have a Beck Suicide Scale score of 5 or higher for the 1-week period prior to admission,
4. are fluent in English,
5. are able to be reached reliably by telephone.

Exclusion Criteria:

1. substantially cognitively impaired (according to the Mini-Cog),
2. unable to provide informed consent for any reason (including incompetency),
3. determined by the patient's attending psychiatrist that peer mentorship is not appropriate due to unstable psychosis, cognitive disorder, or severe personality disorder,
4. already receiving or intending to receive peer mentorship (i.e., sponsor from Alcoholics Anonymous) or group-based peer support on a biweekly or more frequent basis,
5. residing more than 50 miles from any peer mentor,
6. planning to be discharged to another inpatient or residential facility, or
7. receiving electroconvulsive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pfeiffer, MD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - University of Michigan Inpatient Psychiatry Unit, Ann Arbor, Michigan
  - Henry Ford Kingswood Hospital, Ferndale, Michigan
  - Henry Ford Macomb Hospital, Mount Clemens, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pfeiffer PN, Abraham KM, Lapidos A, Vega E, Jagusch J, Garlick J, Pasiak S, Ganoczy D, Kim HM, Ahmedani B, Ilgen M, King C. Peer Support Intervention for Suicide Prevention Among High-Risk Adults in Michigan: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2510808. doi: 10.1001/jamanetworkopen.2025.10808. PMID 40434775
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617

RESULTS

PARTICIPANT FLOW:
Groups:
- Peer Mentorship Intervention (PREVAIL): A Peer Specialist will be making regular follow-up contact with study participants in the community or by telephone for 3 months following hospital discharge. Peer mentorship interactions will include a series of manualized, semi-structured conversations developed by the study team and will address protective factors such as hope and belongingness. PREVAIL arm participants will also receive Enhanced Usual Care (EUC).
  Peer mentorship: The PREVAIL intervention will be delivered by a Certified Peer Support Specialist (CPSS) or Peer Recovery Coach. Participants will select a Peer to work with based on brief personal descriptions. Sessions may occur in-person (public place, the participant's home, or a research clinic space) or remotely (phone or video call). The first meeting will occur while the participant is hospitalized, and subsequent sessions will be scheduled per the participant's preferences, with a suggested frequency of twice weekly for weeks 1-2, weekly for weeks 3-8, and every other week for the last month. Sessions will last 1 hour on average and will consist of semi-structured conversations focused on protective factors such as hope, safety planning, and coping skills. Session structure and content are intentionally flexible to allow for general supportive listening, validation, sharing, and genuineness in the relationship, thereby increasing acceptability and implicit belongingness.
- Enhanced Usual Care (EUC): The EUC condition will consist of a "caring message" from the study team via e-mail or text message (based on the participant's preference) 24-72 hours after discharge. An example message is, "We hope things are going well for you since you left the hospital. If you wish to reply, we'd be glad to hear from you." A list of local mental health resources will be available if participants reply and during the 3 and 6-month follow-up assessments. The EUC condition is modeled on prior studies of caring letters and brief contacts by health professionals after suicidal crisis and national recommendations to provide post-crisis follow-up contacts.
  Enhanced Usual Care: The EUC condition will consist of a "caring message" from the study team via e-mail or text message (based on the participant's preference) 24-72 hours after discharge. An example message is, "We hope things are going well for you since you left the hospital. If you wish to reply, we'd be glad to hear from you". A list of local mental health resources will be available if participants reply and during the 3 and 6-month follow-up assessments. The EUC condition is modeled on prior studies of caring letters and brief contacts by health professionals after suicidal crisis and national recommendations to provide post-crisis follow-up contacts.
Period: Overall Study
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Started | 229 | 226
Completed | 141 | 142
Not Completed | 88 | 84

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC) | Total
Number analyzed (Participants) | 229 | 226 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.40 (14.04) | 31.61 (13.45) | 32.01 (13.74)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 78 | 76 | 154
  Gender: Female | 134 | 139 | 273
  Gender: Other | 17 | 11 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 15 | 23
  Not Hispanic or Latino | 220 | 211 | 431
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 7 | 8 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 40 | 77
  White | 167 | 162 | 329
  More than one race | 16 | 13 | 29
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 229 | 226 | 455
Suicide attempts, as measured by the Columbia Suicide Severity Rating Scale (CSSRS) [Count of Participants; unit: Participants] — Number of participants reporting any suicide attempt, as reported on the Columbia Suicide Severity Rating Scale (CSSRS). The definition of suicide attempt for the primary outcome will consist of any actual suicide attempt, aborted suicide attempt, or interrupted suicide attempt reported on the CSSR-S.
  Participants | 197 | 210 | 407
Suicidal ideation (past week), as measured by the Beck Suicide Scale (BSS) [Mean (Standard Deviation); unit: units on a scale] — Patient's suicidal ideation during the week prior to inpatient psychiatric admission, as measured by the Beck Scale for Suicidal Ideation (BSS). The BSS is a 19-item (5 screening items are first administered to determine whether the remaining items are administered) self-report scale that assesses thoughts, plans and intent to commit suicide. All 19 items are rated on a three-point scale (0 to 2). Total scores could range from 0 to 38. No specific cut-off scores exist to classify severity. Higher scores mean a worse outcome (greater suicide risk).
  units on a scale | 22.00 (7.89) | 22.70 (7.03) | 22.35 (7.47)
Self efficacy to avoid suicidal action (measured by the Self Efficacy to Avoid Suicidal Action Scale [Mean (Standard Deviation); unit: units on a scale] — Participants' sense of self-efficacy to avoid suicidal action, as measured by the 6-item Self Efficacy to Avoid Suicidal Action Scale (SEASA). To indicate level of confidence, respondents rate each item on a 9-point scale (where 0=very uncertain and 9=very certain). Scores range between 0 and 54; lower scores are associated with worse outcomes (a higher incidence and greater severity of suicide attempts).
  units on a scale | 31.77 (14.15) | 29.30 (13.59) | 30.54 (13.91)
Depression, as measured by the Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ-9) is a 9-item, self-report survey which assesses frequency of depression symptoms over the past 2 weeks on a 4-item response scale (where 0 = "Not at all" and 3 = "Nearly every day"). Scores range between 0 and 27, with high scores indicating worse outcomes (more severe depression) Population: Counts of participants analyzed differ from the overall number of participants because some participants did not answer all survey questions.
  units on a scale
    number analyzed (Participants) | 228 | 226 | 454
    (all) | 18.33 (6.57) | 18.33 (5.81) | 18.33 (6.19)
Hope, as measured by the State Hope Scale (SHS) [Mean (Standard Deviation); unit: units on a scale] — The State Hope Scale (SHS) is a 6-item, self-report measure that assesses hopeful thinking along two sub-scales reflecting respondents' personal capacity for change (agency) and knowledge regarding how to achieve change (pathways). Total scores range from 6 to 48. Higher scores indicated better outcomes (greater hope). Population: The number analyzed differs from the overall number of participants because some participants did not respond to all survey questions.
  units on a scale
    number analyzed (Participants) | 228 | 226 | 454
    (all) | 27.34 (10.94) | 25.58 (10.29) | 26.47 (10.65)
Burdensomeness, as measured by the perceived burdensomeness subscale of the Interpersonal Needs Ques [Mean (Standard Deviation); unit: units on a scale] — The Interpersonal Needs Questionnaire (INQ-10) is a 10-item, self-report measure of perceived burdensomeness and thwarted belongingness. The perceived burdensomeness subscale of the INQ-10 consists of 4 items; scores range from 4 to 28, with higher scores indicating worse outcomes (lower perceived belongingness). Population: The number analyzed differs from the overall number of participants because some participants did not respond to all survey questions.
  units on a scale
    number analyzed (Participants) | 228 | 226 | 454
    (all) | 16.01 (8.93) | 16.19 (8.50) | 16.10 (8.71)
Thwarted Belongingness, as Measured by the Thwarted Belongingness Subscale of the INQ-10 [Mean (Standard Deviation); unit: units on a scale] — The Interpersonal Needs Questionnaire (INQ-10) is a 10-item, self-report measure of perceived burdensomeness and thwarted belongingness. The thwarted belongingness subscale of the INQ-10 consists of 6 items; scores range from 5 to 35, with higher scores indicating worse outcomes (greater thwarted belongingness). Population: The number analyzed differs from the overall number of participants because some participants did not respond to all survey questions.
  units on a scale
    number analyzed (Participants) | 228 | 226 | 454
    (all) | 22.33 (7.14) | 23.04 (6.88) | 22.69 (7.01)
Utilization of Health Care Services (Measured by the Adapted Health Services Inventory) [Count of Participants; unit: Participants] — Count of participants who self-reported utilizing any mental health care services on an adapted version of the Health Services Inventory.
  Participants | 194 | 182 | 376
Hopelessness (Measured by the Beck Hopelessness Scale (BHS)) [Mean (Standard Deviation); unit: units on a scale] — Measure of patients' negative attitudes about the future and will be the primary measure of hopelessness. The BHS consists of 20 true-false statements that measure the degree of pessimism and negativity about the future. Summed scores range from 0 to 20. Scores provide a measure of the severity of self-reported hopelessness: 0-3 minimal, 4-8 mild, 9-14 moderate, and 15-20 severe. Population: The number analyzed differs from the overall number of participants because some participants did not respond to all survey questions.
  units on a scale
    number analyzed (Participants) | 228 | 226 | 454
    (all) | 8.42 (5.92) | 9.81 (6.06) | 9.11 (6.03)
Perceived Rejection (Measured by the NIH Toolbox Adult Social Relationship Scales (ASRS)) [Mean (Standard Deviation); unit: units on a scale] — The Adult Toolbox Social Relationship Scales measures social relationship concepts including social support, companionship, and social distress. The perceived rejection subscale consists of 8 items rated on a 5-point Likert scale. Scores range from 8 to 40; higher scores indicate worse outcomes (greater loneliness). Population: The number analyzed differs from the overall number of participants because some participants did not respond to all survey questions.
  units on a scale
    number analyzed (Participants) | 228 | 226 | 454
    (all) | 22.35 (8.13) | 22.78 (7.68) | 22.56 (7.90)
Perceived Emotional Support (measured by the NIH Toolbox Adult Social Relationship Scales (ASRS)) [Mean (Standard Deviation); unit: units on a scale] — The Adult Toolbox Social Relationship Scales measures social relationship concepts including social support, companionship, and social distress. The Emotional Support subscale consists of 8 items rated on a 5-point Likert scale. Scores range from 8 to 40; higher scores indicate better outcomes (greater perceived emotional support). Population: The number analyzed differs from the overall number of participants because some participants did not respond to all survey questions.
  units on a scale
    number analyzed (Participants) | 228 | 226 | 454
    (all) | 27.51 (8.74) | 27.20 (7.93) | 27.35 (8.34)
Perceived Instrumental Support (measured by the NIH Toolbox Adult Social Relationship Scales (ASRS)) [Mean (Standard Deviation); unit: units on a scale] — The Adult Toolbox Social Relationship Scales measures social relationship concepts including social support, companionship, and social distress. The Instrumental Support subscale consists of 8 items rated on a 5-point Likert scale. Scores range from 8 to 40; higher scores indicate better outcomes (greater perceived instrumental support). Population: The number analyzed differs from the overall number of participants because some participants did not respond to all survey questions.
  units on a scale
    number analyzed (Participants) | 228 | 226 | 454
    (all) | 25.83 (9.78) | 26.12 (9.41) | 25.97 (9.59)
Perceived Friendship (Measured by the NIH Toolbox Adult Social Relationship Scales (ASRS)) [Mean (Standard Deviation); unit: units on a scale] — The Adult Toolbox Social Relationship Scales measures social relationship concepts including social support, companionship, and social distress. The Friendship subscale consists of 8 items rated on a 5-point Likert scale. Scores range from 8 to 40; higher scores indicate better outcomes (greater perceived friendship). Population: The number analyzed differs from the overall number of participants because some participants did not respond to all survey questions.
  units on a scale
    number analyzed (Participants) | 228 | 226 | 454
    (all) | 21.41 (8.09) | 22.57 (8.35) | 21.99 (8.23)
Loneliness (measured by the NIH Toolbox Adult Social Relationship Scales (ASRS)) [Mean (Standard Deviation); unit: units on a scale] — The Adult Toolbox Social Relationship Scales measures social relationship concepts including social support, companionship, and social distress. The Loneliness subscale consists of 5 items rated on a 5-point Likert scale. Scores range from 5 to 25; higher scores indicate worse outcomes (greater loneliness).
  units on a scale | 17.74 (4.67) | 17.85 (4.70) | 17.80 (4.68)
Highest level of education [Count of Participants; unit: Participants]
  8th grade or less | 1 | 3 | 4
  Some high school | 19 | 11 | 30
  High school graduate/GED | 53 | 49 | 102
  Some college | 98 | 98 | 196
  College graduate | 44 | 45 | 89
  Advanced degree | 14 | 20 | 34
Marital Status [Count of Participants; unit: Participants]
  Married | 45 | 35 | 80
  Divorced/separated | 30 | 29 | 59
  Widowed | 2 | 9 | 11
  Never married | 137 | 134 | 271
  Living together, not married | 15 | 19 | 34
Occupation [Count of Participants; unit: Participants] — Participants could select more than one occupation if applicable.
  Participants
    Homemaker/Caregiver | 11 | 15 | 26
    Retired | 10 | 9 | 19
    Working part-time | 45 | 51 | 96
    Working full-time | 71 | 73 | 144
    Volunteering full-time | 1 | 0 | 1
    Volunteering part-time | 2 | 5 | 7
    Unemployed or on disability | 58 | 57 | 115
    Student | 67 | 62 | 129
    Missing/declined to answer | 2 | 1 | 3
Income (annual) [Count of Participants; unit: Participants]
  Under $5,000 | 56 | 60 | 116
  $5,000 - $14,999 | 48 | 48 | 96
  $15,000 - $24,999 | 41 | 34 | 75
  $25,000 - $49,000 | 43 | 44 | 87
  $50,000 - $74,999 | 16 | 21 | 37
  $75,000 - $99,999 | 10 | 7 | 17
  $100,000 or more | 9 | 8 | 17
  Missing/declined to answer | 6 | 4 | 10
Living Situation [Count of Participants; unit: Participants] — Participants could select more than one option if applicable.
  Participants
    Lives with spouse or partner | 65 | 64 | 129
    Lives with parents | 61 | 67 | 128
    Lives with children under age 18 | 39 | 43 | 82
    Lives with other relatives or friends | 61 | 47 | 108
    Lives with others, but not friends or relatives | 7 | 16 | 23
    Lives alone | 32 | 41 | 73
    Homeless or between housing arrangements | 22 | 14 | 36
Quality of Life (Measured by the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form [Mean (Standard Deviation); unit: units on a scale] — Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) consists of 14 items, assesses satisfaction with a variety of life domains such as physical health, work, and social relationships. The scoring of the Q-LES-Q-SF involves summing only the first 14 items to yield a raw total score. The last two items are not included in the total score but are standalone items. The raw total score ranges from 14 to 70. Higher level of enjoyment and satisfaction with life are reflected in higher scores. Population: Counts of participants analyzed differ from the overall number of participants because some participants did not answer all survey questions.
  units on a scale
    number analyzed (Participants) | 228 | 226 | 454
    (all) | 39.18 (10.30) | 38.80 (9.84) | 38.99 (10.06)
Physical Health (Measured by the SF-12) [Mean (Standard Deviation); unit: units on a scale] — The SF-12 covers domains including: (1) physical functioning; (2) role-physical; (3) bodily pain; (4) general health; (5) vitality; (6) social functioning; (7) role emotional; and (8) mental health. Physical Health Composite Score (PCS) is computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Population: Counts of participants analyzed differ from the overall number of participants because some participants did not answer all survey questions.
  units on a scale
    number analyzed (Participants) | 227 | 222 | 449
    (all) | 51.71 (12.24) | 51.36 (13.18) | 51.54 (12.70)
Mental Health (measured by the SF-12) [Mean (Standard Deviation); unit: units on a scale] — The SF-12 covers domains including: (1) physical functioning; (2) role-physical; (3) bodily pain; (4) general health; (5) vitality; (6) social functioning; (7) role emotional; and (8) mental health. Mental Health Composite Score (MCS) is computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Population: Counts of participants analyzed differ from the overall number of participants because some participants did not answer all survey questions.
  units on a scale
    number analyzed (Participants) | 227 | 222 | 449
    (all) | 23.48 (10.68) | 23.76 (11.00) | 23.62 (10.83)
Perceived Social Support (Measured by the Multidimensional Scale of Perceived Social Support (MDPSS) [Mean (Standard Deviation); unit: units on a scale] — The Multidimensional Scale of Perceived Social Support (MDPSS) contains 12 Likert scale items with three subscales to address different sources of support: family, friends, and significant other. Mean scores under 2.9 are considered low support, mean scores 3-5 are considered moderate, and 5.1-7 are considered high. The family and friend support subscales score ranges from 1-7. Total item mean is the mean of all single item means and ranges from 1-7. Higher scores indicate greater social support. Population: Counts of participants analyzed differ from the overall number of participants because some participants did not answer all survey questions.
  units on a scale
    Total item mean: number analyzed (Participants) | 227 | 226 | 453
    Total item mean | 4.70 (1.59) | 4.59 (1.39) | 4.64 (1.59)
    Family subscale | 4.43 (1.96) | 4.07 (1.79) | 4.25 (1.88)
    Friend subscale | 4.57 (1.95) | 4.80 (1.67) | 4.68 (1.81)
Perceived Meaning in Life, as Measured by the Meaning in Life Questionnaire (MLQ) [Mean (Standard Deviation); unit: units on a scale] — The Meaning in Life Questionnaire (MLQ) consists of 10 items measured on a 7-point likert scale ranging from absolutely true to absolutely not true. The measure consists of two subscales - presence of meaning and search for meaning. Subscale scores range from 5 to 35; higher scores indicate better outcomes (greater meaning). Population: Counts of participants analyzed differ from the overall number of participants because some participants did not answer all survey questions.
  units on a scale
    Presence subscale: number analyzed (Participants) | 228 | 226 | 454
    Presence subscale | 18.41 (8.44) | 17.35 (8.07) | 17.88 (8.27)
    Searching subscale: number analyzed (Participants) | 227 | 226 | 453
    Searching subscale | 25.80 (7.68) | 25.46 (7.15) | 25.63 (7.41)

OUTCOME MEASURES:

1. Primary Outcome: Suicide Attempts, as Measured by the Columbia Suicide Severity Rating Scale (CSSRS)
Description: Number of participants reporting any suicide attempt, as reported on the Columbia Suicide Severity Rating Scale (CSSRS). The definition of suicide attempt for the primary outcome will consist of any actual suicide attempt, aborted suicide attempt, or interrupted suicide attempt reported on the CSSR-S.
Time Frame: 3 months, 6 months
Population: The number of participant analyzed decreases at the 3- and 6-month time points due to attrition.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 229 | 226
Participants
  3 Months - count of participants with any suicide attempt (actual, interrupted, or aborted): number analyzed (Participants) | 142 | 151
  3 Months - count of participants with any suicide attempt (actual, interrupted, or aborted) | 13 | 17
  6 Months - count of participants with any suicide attempt (actual, interrupted, or aborted): number analyzed (Participants) | 161 | 163
  6 Months - count of participants with any suicide attempt (actual, interrupted, or aborted) | 24 | 28
Statistical Analysis 1: Comparison: Peer Mentorship Intervention (PREVAIL) vs Enhanced Usual Care (EUC); Test type: Other; p = 0.58, Chi-squared

2. Primary Outcome: Suicidal Ideation (Current), as Measured by the Beck Suicide Scale (BSS)
Description: Patient's current suicidal ideation as measured by the Beck Scale for Suicidal Ideation (BSS). The BSS is a 19-item (5 screening items are first administered to determine whether the remaining items are administered) self-report scale that assesses thoughts, plans and intent to commit suicide. All 19 items are rated on a three-point scale (0 to 2). Total scores could range from 0 to 38. No specific cut-off scores exist to classify severity. Higher scores mean a worse outcome (greater suicide risk).
Time Frame: 3 months, 6 months
Population: The number of participant analyzed decreases at the 3- and 6-month time points due to attrition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 229 | 226
units on a scale
  3 Months: number analyzed (Participants) | 149 | 158
  3 Months | 4.15 (6.55) | 4.37 (6.80)
  6 Months: number analyzed (Participants) | 141 | 142
  6 Months | 4.86 (7.32) | 4.25 (6.62)
Statistical Analysis 1: Comparison: Peer Mentorship Intervention (PREVAIL) vs Enhanced Usual Care (EUC); Test type: Other; p = 0.46, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Suicide Attempts (Measured by the Medical Record)
Description: Count of participants with any suicide attempt as notated in the patient's electronic medical record. The definition of suicide attempt for the primary outcome will consist of any actual suicide attempt, aborted suicide attempt, or interrupted suicide attempt.
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 229 | 226
Participants | 11 | 9
Statistical Analysis 1: Comparison: Peer Mentorship Intervention (PREVAIL) vs Enhanced Usual Care (EUC); Test type: Other; p = 0.18, Chi-squared

4. Secondary Outcome: Self Efficacy to Avoid Suicidal Action (Measured by the Self Efficacy to Avoid Suicidal Action Scale)
Description: Participants' sense of self-efficacy to avoid suicidal action, as measured by the 6-item Self Efficacy to Avoid Suicidal Action Scale (SEASA). To indicate level of confidence, respondents rate each item on a 9-point scale (where 0=very uncertain and 9=very certain). Scores range between 0 and 54; lower scores are associated with worse outcomes (a higher incidence and greater severity of suicide attempts).
Time Frame: 3 months, 6 months
Population: Number of participants analyzed decreases at 3- and 6-month time points due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 229 | 226
score on a scale
  3 Months: number analyzed (Participants) | 149 | 158
  3 Months | 36.12 (13.35) | 34.64 (13.04)
  6 months: number analyzed (Participants) | 141 | 142
  6 months | 37.06 (11.69) | 35.52 (12.03)
Statistical Analysis 1: Comparison: Peer Mentorship Intervention (PREVAIL) vs Enhanced Usual Care (EUC); Test type: Other; p = 0.29, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Suicidal Ideation (Worst-point), as Measured by the Beck Scale for Suicidal Ideation (BSS)
Description: Patient's worst-point suicidal ideation as measured by the Beck Scale for Suicidal Ideation (BSS). The BSS is a 19-item (5 screening items are first administered to determine whether the remaining items are administered) self-report scale that assesses thoughts, plans and intent to commit suicide. All 19 items are rated on a three-point scale (0 to 2). Total scores could range from 0 to 38. No specific cut-off scores exist to classify severity. Higher scores mean a worse outcome (greater suicide risk).
Time Frame: 3 months, 6 months
Population: Number of participants analyzed decreases at 3- and 6-month time points due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 229 | 226
score on a scale
  3-Months: number analyzed (Participants) | 149 | 158
  3-Months | 10.66 (10.50) | 10.53 (9.92)
  6-Months: number analyzed (Participants) | 141 | 142
  6-Months | 7.76 (9.14) | 8.68 (9.30)
Statistical Analysis 1: Comparison: Peer Mentorship Intervention (PREVAIL) vs Enhanced Usual Care (EUC); Test type: Other; p = 0.35, Wilcoxon (Mann-Whitney)

6. Other Pre Specified Outcome: Depression, as Measured by the Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) is a 9-item, self-report survey which assesses frequency of depression symptoms over the past 2 weeks on a 4-item response scale (where 0 = "Not at all" and 3 = "Nearly every day"). Scores range between 0 and 27, with high scores indicating worse outcomes (more severe depression)
Time Frame: 3 months, 6 months
Population: Number of participants analyzed decreases at 3- and 6-month time points due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 229 | 226
score on a scale
  3-Months: number analyzed (Participants) | 149 | 158
  3-Months | 10.83 (6.86) | 10.75 (6.87)
  6-Months: number analyzed (Participants) | 141 | 142
  6-Months | 11.56 (7.27) | 10.84 (6.71)

7. Other Pre Specified Outcome: Hope, as Measured by the State Hope Scale (SHS)
Description: The State Hope Scale (SHS) is a 6-item, self-report measure that assesses hopeful thinking along two sub-scales reflecting respondents' personal capacity for change (agency) and knowledge regarding how to achieve change (pathways). Total scores range from 6 to 48. Higher scores indicated better outcomes (greater hope).
Time Frame: 3-months
Population: Number of participants analyzed decreases at 3- and 6-month time points due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 229 | 226
score on a scale | 32.12 (10.37) | 30.57 (9.77)

8. Other Pre Specified Outcome: Burdensomeness, as Measured by the Perceived Burdensomeness Subscale of the Interpersonal Needs Questionnaire (INQ-10)
Description: The Interpersonal Needs Questionnaire (INQ-10) is a 10-item, self-report measure of perceived burdensomeness and thwarted belongingness. The perceived burdensomeness subscale of the INQ-10 consists of 4 items; scores range from 4 to 28, with higher scores indicating worse outcomes (greater perceived burdensomeness).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale | 12.03 (8.21) | 11.87 (7.66)

9. Other Pre Specified Outcome: Perceived Emotional Support (Measured by the NIH Toolbox Adult Social Relationship Scales (ASRS))
Description: The Adult Toolbox Social Relationship Scales measures social relationship concepts including social support, companionship, and social distress. The Emotional Support subscale consists of 8 items rated on a 5-point Likert scale. Scores range from 8 to 40; higher scores indicate better outcomes (greater perceived emotional support).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale | 31.33 (7.85) | 30.97 (7.25)

10. Other Pre Specified Outcome: Perceived Instrumental Support (Measured by the NIH Toolbox Adult Social Relationship Scales (ASRS))
Description: The Adult Toolbox Social Relationship Scales measures social relationship concepts including social support, companionship, and social distress. The Instrumental Support subscale consists of 8 items rated on a 5-point Likert scale. Scores range from 8 to 40; higher scores indicate better outcomes (greater perceived instrumental support).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale | 28.46 (9.67) | 28.90 (9.07)

11. Other Pre Specified Outcome: Perceived Friendship (Measured by the NIH Toolbox Adult Social Relationship Scales (ASRS))
Description: The Adult Toolbox Social Relationship Scales measures social relationship concepts including social support, companionship, and social distress. The Friendship subscale consists of 8 items rated on a 5-point Likert scale. Scores range from 8 to 40; higher scores indicate better outcomes (greater perceived friendship).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale | 24.26 (8.96) | 24.69 (8.37)

12. Other Pre Specified Outcome: Loneliness (Measured by the NIH Toolbox Adult Social Relationship Scales (ASRS))
Description: The Adult Toolbox Social Relationship Scales measures social relationship concepts including social support, companionship, and social distress. The Loneliness subscale consists of 5 items rated on a 5-point Likert scale. Scores range from 5 to 25; higher scores indicate worse outcomes (greater loneliness).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale | 15.19 (6.03) | 15.02 (5.30)

13. Other Pre Specified Outcome: Perceived Rejection (Measured by the NIH Toolbox Adult Social Relationship Scales (ASRS))
Description: The Adult Toolbox Social Relationship Scales measures social relationship concepts including social support, companionship, and social distress. The perceived rejection subscale consists of 8 items rated on a 5-point Likert scale. Scores range from 8 to 40; higher scores indicate worse outcomes (greater loneliness).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale | 18.43 (8.53) | 19.14 (8.22)

14. Other Pre Specified Outcome: Quality of Life (Measured by the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF))
Description: Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) consists of 14 items, assesses satisfaction with a variety of life domains such as physical health, work, and social relationships. The scoring of the Q-LES-Q-SF involves summing only the first 14 items to yield a raw total score. The last two items are not included in the total score but are standalone items. The raw total score ranges from 14 to 70. Higher level of enjoyment and satisfaction with life are reflected in higher scores.
Time Frame: 3 months, 6 months
Population: The number of participants analyzed decreases at 6-months due to attrition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale
  3-Months | 46.41 (11.42) | 45.82 (10.15)
  6-Months: number analyzed (Participants) | 141 | 142
  6-Months | 46.05 (11.98) | 46.46 (10.81)

15. Other Pre Specified Outcome: Functional Status (Measured by the SF-12)
Description: The SF-12 covers domains including: (1) physical functioning; (2) role-physical; (3) bodily pain; (4) general health; (5) vitality; (6) social functioning; (7) role emotional; and (8) mental health. Summary scores are calculated by summing factor-weighted scores across all 8 subscales, with factor weights derived from a US-based general population sample. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: 3 months, 6 months
Population: Number of participants analyzed decreases at 6-months due to attrition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale
  3-Months | 48.60 (13.28) | 48.86 (12.72)
  6-Months: number analyzed (Participants) | 141 | 142
  6-Months | 49.18 (12.39) | 48.19 (13.70)

16. Other Pre Specified Outcome: Hopelessness (Measured by the Beck Hopelessness Scale (BHS))
Description: Measure of patients' negative attitudes about the future and will be the primary measure of hopelessness. The BHS consists of 20 true-false statements that measure the degree of pessimism and negativity about the future. Summed scores range from 0 to 20. Scores provide a measure of the severity of self-reported hopelessness: 0-3 minimal, 4-8 mild, 9-14 moderate, and 15-20 severe.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale | 6.27 (5.56) | 6.51 (5.30)

17. Other Pre Specified Outcome: Perceived Social Support (Measured by the Multidimensional Scale of Perceived Social Support (MDPSS))
Description: The Multidimensional Scale of Perceived Social Support (MDPSS) contains 12 Likert scale items with three subscales to address different sources of support: family, friends, and significant other. Total scores are an average (mean) of the subscale scores. Mean scores under 2.9 are considered low support, mean scores 3-5 are considered moderate, and 5.1-7 are considered high. Scores range from 1-7, with 1 representing lowest support and 7 representing highest support.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale | 5.08 (1.59) | 4.91 (1.43)

18. Other Pre Specified Outcome: Self-reported Utilization of Health Care Services, as Measured by the Adapted Health Services Inventory
Description: Count of participants who self-reported utilizing any mental health care services.
Time Frame: 3 months, 6 months
Population: Number of participants analyzed decreases at 6-months due to attrition.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
Participants
  3-Months: number analyzed (Participants) | 138 | 146
  3-Months | 109 | 119
  6-Months: number analyzed (Participants) | 134 | 133
  6-Months | 86 | 98

19. Other Pre Specified Outcome: Medication Adherence, as Measured by the Single-Item Self Rating (SISR) Scale for Medication Adherence
Description: Single item that ask patients' ability to take their medications as their doctor prescribed them, rated on a 6-point scale from 1 = "Excellent" to 6 = "Very Poor," such that higher scores indicate worse outcomes (poorer adherence with taking medications as prescribed).
Time Frame: 3 months, 6 months
Population: Number of participants analyzed is lower at 6-months due to attrition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale
  3-Months | 2.23 (1.53) | 2.16 (1.40)
  6-Months: number analyzed (Participants) | 141 | 142
  6-Months | 2.50 (1.59) | 2.29 (1.32)

20. Other Pre Specified Outcome: Perceived Meaning in Life, as Measured by the Meaning in Life Questionnaire (MLQ)
Description: The Meaning in Life Questionnaire (MLQ) consists of 10 items measured on a 7-point likert scale ranging from absolutely true to absolutely not true. The measure consists of two subscales: presence of meaning and search for meaning. Subscale scores range from 5 to 35; higher scores indicated better outcomes (greater meaning).
Time Frame: 3 months, 6 months
Population: Number of participants analyzed decreases at 6-months due to attrition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale
  Presence subscale: 3-Months | 21.96 (8.89) | 20.45 (8.51)
  Presence subscale: 6-Months: number analyzed (Participants) | 141 | 142
  Presence subscale: 6-Months | 21.48 (8.73) | 19.90 (8.47)
  Searching subscale: 3-Months | 25.80 (7.38) | 25.15 (7.00)
  Searching subscale: 6-Months | 25.73 (7.33) | 25.02 (7.01)

21. Other Pre Specified Outcome: Worst Suicidal Ideation in Past 3 Months (Measured by the Beck Suicide Scale (BSS))
Description: Patient's worst suicidal ideation in the previous 3-month time period as measured by the Beck Suicide Scale (BSS). The BSS is a self-report 19-item scale preceded by five screening items. The BSS and its screening items assess thoughts, plans and intent to commit suicide. All 24 items are rated on a three-point scale (0 to 2). Total scores could range from 0 to 38 (if the screening items are included). No specific cut-off scores exist to classify severity. Increasing scores reflect greater suicide risk.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale | 10.66 (10.50) | 10.53 (9.92)

22. Other Pre Specified Outcome: Worst Suicidal Ideation in Past 3 Months (Measured by the Beck Suicide Scale (BSS))
Description: as for outcome 21
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 141 | 142
units on a scale | 7.76 (9.14) | 8.68 (9.30)

23. Other Pre Specified Outcome: Thwarted Belongingness, as Measured by the Thwarted Belongingness Subscale of the Interpersonal Needs Questionnaire (INQ-10)
Description: The Interpersonal Needs Questionnaire (INQ-10) is a 10-item, self-report measure of perceived burdensomeness and thwarted belongingness. The thwarted belongingness subscale of the INQ-10 consists of 6 items; scores range from 5 to 35, with higher scores indicating worse outcomes (greater thwarted belongingness).
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 149 | 158
units on a scale | 18.92 (7.85) | 19.51 (8.04)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Peer Mentorship Intervention (PREVAIL) | Enhanced Usual Care (EUC)
All-Cause Mortality (participants affected / at risk) | 2/229 | 2/226
Serious Adverse Events (participants affected / at risk) | 51/229 | 55/226
Other Adverse Events (participants affected / at risk) | 0/229 | 0/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Mentorship Intervention (PREVAIL) (N=229) | Enhanced Usual Care (EUC) (N=226)
Medically serious suicide attempt (Psychiatric disorders) | 3 (3) | 2 (2) — Suicide attempt requiring medical hospitalization.
Psychiatric hospitalization due to suicidal intent or behavior (Psychiatric disorders) | 27 (35) | 29 (38)
Psychiatric hospitalization for a reason other than suicide risk (Psychiatric disorders) | 4 (4) | 3 (3)
Psychiatric Emergency Department visit without hospitalization (Psychiatric disorders) | 10 (14) | 9 (9)
Homicidal behavior (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt without medical attention (Psychiatric disorders) | 6 (12) | 12 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT03373916/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT03373916/ICF_001.pdf